CLINICAL TRIAL: NCT05243147
Title: Clinical Control Study of Application of Nasal Stent and Merocel Sponge After Nasal Septoplasty
Brief Title: Design and Application of Nasal Stents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUTH-NS
Record Dates: First submitted 2021-12-28; First posted 2022-02-16 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2022-12

CONDITIONS: Nasal Septum; Deviation, Congenital

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nasal stents (Experimental): using nasal stents after septoplasty
  Interventions: Device: nasal stents
- merocel (Other): using merocel as nasal packing after septoplasty
  Interventions: Device: merocel

INTERVENTIONS:
Device: nasal stents — using nasal stents after septoplasty
  Arms: nasal stents
Device: merocel — using merocel after septoplasty
  Arms: merocel

SUMMARY:
Comparative study of nasal stents and nasal packing in patients undergoing septoplasty

DETAILED DESCRIPTION:
To investigate the safety and effectiveness of nasal stent in clinical application by comparing and observing the clinical effect and comfort of nasal stent and merocel sponge applied in nasal septoplasty. Methods: patients with nasal septal deviation were selected and randomly divided into nasal stent group (experimental group) and merocel sponge group (control group) according to the packing method. The hemostasis effect, comfort and complications of the two groups were compared during the packing period.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily participate in the experiment and sign the informed consent;
2. Age range from 18 to 70 years old, gender unlimited;
3. With nasal congestion as the chief complaint, CT of sinus suggested deviation of nasal septum with indications of surgery (deviation of nasal septum affects breathing and nasal congestion is serious; High nasal septum deviation affects sinus drainage or causes reflex headache; Nasal septum spine often causes nasal bleeding; Nasal septum deviation affects eustachian tube function);
4. No history of respiratory tract infection and nasal decongestant use within 1 month before the visit;
5. No other treatment was used;
6. ASA grade 1~2;
7. Able to communicate well with researchers and follow the requirements of the experiment.

Exclusion Criteria:

1. There are acute and chronic rhinosinusitis, nasal polyps, benign and malignant tumors and other nasal diseases;
2. History of craniocerebral and nasal surgery;
3. The results of preoperative coagulation function test exceeded 20% of the upper limit of normal value;
4. Patients known to be allergic to test instrument materials;
5. Pregnant or lactating women;
6. Other organoplastic or functional diseases complicated by the subjects limited their participation in the study and could not comply with the follow-up or affect the scientific integrity of the study;
7. Participants who have participated in other clinical trials within the last 1 month;
8. Participants considered unsuitable for this clinical trial for other reasons.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Effective rate of packing | 2days after operation
  (1) In the period of nasal tamponade and after the removal of the tamponade instrument (48 h ± 1 h after surgery), the nasal bleeding score was ≤ 2 points; (2) 48 h ± 1 h after the completion of nasal tamponade, the overall discomfort score ≤ 7 points; (3) No septal hematoma and nasal adhesions were confirmed by nasal endoscopy at 30 days ± 5 days after the operation. Nasal tamponade is considered effective when the above 3 criteria are met.

SECONDARY OUTCOMES:
visual analog scale（VAS）of comfort | 2days after operation
  including nasal congestion, nasal pain, headache, itchy nose sneezing, watery tears, runny nose, nasal reflux, facial swelling, difficulty swallowing, sleep disturbance, dry mouth, and general discomfort. The severity of each symptom was graded using the visual analog scale (VAS) of 0 (none) to10 (unbearable)
security | 30days after operation
  The incidence of complications and adverse events were used as safety evaluation indexes

CONTACTS AND LOCATIONS:
Overall Officials: Junxiu Liu, Principal Investigator — Peking University Third Hosptial
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No